CLINICAL TRIAL: NCT05144464
Title: A Clinical Trial to Assess Immunogencity and Safety of 2 Doses of an Inactivated Quadrivalent Influenza Vaccine in Chinese Children Aged 3 to 8 Years
Brief Title: A Clinical Trial of an Inactivated Quadrivalent Influenza Vaccine in Chinese Children Aged 3 to 8 Years
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Jiangsu Jindike Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT122
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Safety, Immunogenicity, Quadrivalent influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Subjects received 2 doses of an inactivated quadrivalent influenza vaccine, 4 weeks apart. Blood samples were obtained from children at 3 time points-before receipt of dose 1, 4 weeks after receipt of dose 1 and before dose 2, and 4 weeks after dose 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quadrivalent influenza vaccine (Experimental): Subjects received 2 doses of 0.5 mL of quadrivalent influenza vaccine, 4 weeks apart. Each 0.5-ml dose contained 15 μg of hemagglutinin per strain.
  Interventions: Biological: Quadrivalent influenza vaccine

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine — Subjects receive two doses of quadrivalent influenza vaccine administered 4 weeks apart by intramuscular injection

SUMMARY:
Routine annual influenza vaccination is recommended for all persons aged ≥6 months who do not have contraindications. For those aged 6 months through 8 years who have previously received ≥2 total doses of trivalent or quadrivalent influenza vaccine ≥4 weeks apart, they require only 1 dose of influenza vaccine. For those who have not previously received ≥2 doses of trivalent or quadrivalent influenza vaccine, they require 2 dose of influenza vaccine. but the evidence on how to select vaccine doses for quadrivalent influenza vaccine is limited in China. The study is a prospective, open-label comparison of the immunogenicity and reactogenicity of 1 versus 2 doses of an inactivated quadrivalent influenza vaccine in subjects of 3-8 years old with different history of influenza vaccination.

DETAILED DESCRIPTION:
Subjects receive 2 dosed of quadrivalent influenza vaccine 4 weeks apart.

Blood samples were obtained from children at 3 time points-before receipt of dose 1, 4 weeks after receipt of dose 1 and before dose 2, and 4 weeks after dose 2. Hemagglutination inhibition (HAI) antibody titers to the A/H3N2, A/H1N1, and B antigens included in the vaccine were measured at each time point

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-8 years old
* Healthy subjects judged from medical history and clinical examination
* Subjects themselves or their guardians able to understand and sign the informed consent
* Subjects themselves or their guardians can and will comply with the requirements of the protocol
* Subjects have received ≥2 doses of trivalent or quadrivalent infuenza vaccine before enrollment (Doses need not have been received during same or consecutive seasons); Subjects have not received infuenza vaccine before enrollment
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

* Subject who has a medical or family history of any of the following: allergic history, seizure, epilepsy, brain or mental disease
* Subject who is allergic to any ingredient of the vaccine
* Subject with damaged or low immune function which has already been known
* Subject with acute febrile illness or infectious disease
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Thrombocytopenia, blood coagulation disorder or bleeding difficulties with intramuscular injection
* Subject who has serious allergic history
* Subject who developed guillain-Barre syndrome post influenza vaccination
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of influenza vaccine in last 6 month
* Any prior administration of blood products in last 3 months
* Any prior administration of other research medicine/vaccine in last 30 days
* Any prior administration of any attenuated live vaccine in last 14 days
* Any prior administration of subunit or inactivated vaccines in last 7 days, such as pneumococcal vaccine
* Any medical, psychological, social or other condition judged by investigator, that may interfere subject's compliance with the protocol or signature on informed consent for subject's guardian

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2021-09-19 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
the 95% confidence interval (CI) lower limit for Seroconversion Rate (SCR) of Hemagglutination inhibition (HAI) antibodies against each virus strain after 2nd vaccination ≥40% | day 28 after dose 2
  The lowest dilution used in the assay is 1/10. Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and ≥ four-fold increase in post-vaccination titer.
Number of participants with Adverse Reactions (ARs) | 28 days after each vaccination
  Frequency and severity of ARs for 28 days after each vaccination

SECONDARY OUTCOMES:
the 95% CI lower limit for seroprotection rates of HAI antibodies against each virus strain after 2nd vaccination≥70% | day 28 after dose 2
  A seroprotected subject is defined as a vaccinated subject with serum HAI titer≥ 1:40.
Geometric Mean Fold Increase (GMFI) of HAI titer against each virus strain after 2nd vaccination>2.5 | day 28 after dose 2
  Hemagglutination inhibition (HAI) titers were used to calculate post-vaccination geometric mean fold increase (GMFI) against each virus strain
Number of participants with Adverse Events (AEs) | 28 days after each vaccination
  Frequency and severity of AEs for 28 days after each vaccination
Number of participants with Serious Adverse Events (SAE) | 6 months after the last vaccination
  Frequency of SAEs for 6 months after the last vaccination

OTHER OUTCOMES:
Comparision between Seroconversion Rate (SCR) of HAI antibodies against each virus strain post dose 1 and dose 2 | day 28 after receipt of dose 1 and before dose 2, and day 28 after dose 2.
  The lowest dilution used in the assay is 1/10. Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and ≥ four-fold increase in post-vaccination titer.
Comparision between Geometric Mean Titre (GMT) of HAI antibodies against each virus strain post dose 1 and dose 2 | day 28 after receipt of dose 1 and before dose 2, and day 28 after dose 2.
Comparision between seroprotection rates of HAI antibodies against each virus strain post dose 1 and dose 2 | day 28 after receipt of dose 1 and before dose 2, and day 28 after dose 2.
  A seroprotected subject is defined as a vaccinated subject with serum HAI titer≥ 1:40.
Comparision between Geometric Mean Fold Increase (GMFI) of HAI antibodies against each virus strain post dose 1 and dose 2 | day 28 after receipt of dose 1 and before dose 2, and day 28 after dose 2.
  Hemagglutination inhibition (HAI) titers were used to calculate post-vaccination geometric mean fold increase (GMFI) against each virus strain

CONTACTS AND LOCATIONS:
Overall Officials: Fangyue Meng, Master, Principal Investigator — Jiangsu Province Centers for Disease Control and Prevention
Locations (1):
- Pizhou City Center for Disease Control and Prevention, Xuzhou, Jiangsu, China

REFERENCES:
- [Derived] Wen F, Liu S, Zhou L, Zhu Y, Wang W, Wei M, Xu X, Liu Y, Shuai Q, Yu J, Jing P, Li J, Zhu F. Immunogenicity and safety of 1 versus 2 doses of quadrivalent-inactivated influenza vaccine in children aged 3-8 years with or without previous influenza vaccination histories. Hum Vaccin Immunother. 2025 Dec;21(1):2468074. doi: 10.1080/21645515.2025.2468074. Epub 2025 Feb 24. PMID 39993940